CLINICAL TRIAL: NCT05929339
Title: Defining a Pharmacokinetic and Pharmacodynamic Model for Peripheral Analgesia After Intravenous Oxytocin
Brief Title: Defining a PK and PD Model for Peripheral Analgesia After IV Oxytocin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00097699; 1P01NS119159-01A1 (NIH)
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2024-12

CONDITIONS: Acute Pain; Chronic Pain; Healthy Volunteer
Keywords: Acute pain; Chronic Pain; Oxytocin
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: All subjects will receive two 30-minute infusions of oxytocin, 10 IU. The second infusion will be given 30 minutes after the completion of the first infusion. The first 8 subjects report pain at the end of 5 minutes of skin heating at intervals beginning 15 minutes after starting the first infusion. The remaining subjects will be randomized to report pain at the end of 5 minutes of skin heating at intervals beginning at either 10 or 20 minutes after starting the first infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Verbal Pain Score at 10 Minutes (Other): Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 10 minutes after starting the intervention, then every 15 minutes until 115 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Interventions: Drug: Oxytocin
- Verbal Pain Score at 15 Minutes (Other): Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 15 minutes after starting the intervention, then every 15 minutes until 120 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Interventions: Drug: Oxytocin
- Verbal Pain Score at 20 Minutes (Other): Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 20 minutes after starting the intervention, then every 15 minutes until 125 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Intravenous oxytocin
  Other Names: Pitocin

SUMMARY:
The goal of this clinical trial is to learn about oxytocin ( a naturally occurring hormone made in the brain that transmits messages) and the effects it may have on thermal heat pain after intravenous administration. The main question it aims to define is the time course of change in pain score after a 5 minute heating of the skin administered at intervals during and following infusion of intravenous oxytocin in order to create a Pharmacokinetic and a Pharmacodynamic model for oxytocin-induced analgesia.

Participants will be asked to rate thermal heat temperatures before, during and after the intravenous infusion of oxytocin.

DETAILED DESCRIPTION:
The primary objective is to define the time course of change in pain score after a 5 minute heating of the skin applied at intervals during and following infusion of intravenous oxytocin in order to create a Pharmacokinetic and Pharmacodynamic model for oxytocin-induced analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
5. Subjects with current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval.
6. Subjects with past or current history of hyponatremia or at risk for hyponatremia; anyone taking thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, Ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, SSRI's, MAOI, or the recreational drug ecstasy.
7. Subjects with a known latex allergy.
8. Subjects with a pain score rating of 1 or less during the initial training session to a 5 minute heating of 45°C- 47 °Celsius to the lower calf.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Statistical programs in the data analysis will be written in R. The software and anonymized data will be included both as digital supplements in the published papers and will be posted on GitHub under github.com/StevenLShafer. Interested investigators will be able to reproduce the published analyses from these files. Consistent with the posting of software and data to the OpenTCI initiative, the software and de-identified data will be made available with "no strings attached," enabling investigators to freely use the data to inform or supplement additional research without restriction. Data to be made available are oxytocin dose, times of pharmacodynamic measures (relative to the start of dosing), simulated plasma oxytocin concentrations at those times for each subject, and age, weight, and sex for each subject.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available upon publication or upon posting results in ClinicalTrials.gov, whichever comes first, with no expiration.
Access Criteria: These data are freely shared to all and will be posted at the URL below
URL: http://github.com/StevenLShafer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants were recruited from the community from Aug 17, 2023 through October 2, 2024 via IRB-approved advertisements and IRB-approved lists of previous participants who agreed to be contacted for future studies. They were recruited by phone and provided written informed consent at the day of the training visit.
Groups:
- Verbal Pain Score at 10 Minutes: In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 10, 25, 40, 55, 70, 85, 100, 115, and 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the intervention.
- Verbal Pain Score at 15 Minutes: In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 15, 30, 45, 60, 75, 90, 105, 120, and 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the intervention.
- Verbal Pain Score at 20 Minutes: In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 20, 35, 50, 65, 80, 95, 110, 125, and 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the intervention.
Period: Overall Study
Arm/Group | Verbal Pain Score at 10 Minutes | Verbal Pain Score at 15 Minutes | Verbal Pain Score at 20 Minutes
Started | 8 | 8 | 9
Completed | 8 | 8 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Verbal Pain Score at 10 Minutes: In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 10 minutes after starting the intervention, then every 15 minutes until 115 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the intervention.
- Verbal Pain Score at 15 Minutes: In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 15 minutes after starting the intervention, then every 15 minutes until 120 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the intervention.
- Verbal Pain Score at 20 Minutes: In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 20 minutes after starting the intervention, then every 15 minutes until 125 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the intervention.
- Total: Total of all reporting groups
Arm/Group | Verbal Pain Score at 10 Minutes | Verbal Pain Score at 15 Minutes | Verbal Pain Score at 20 Minutes | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (19) | 24 (4) | 42 (21) | 38 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 6 | 8 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 | 25
Verbal pain score at the end of 5 minute skin heating [Mean (Standard Deviation); unit: units on a scale] | 3.9 (0.8) | 3.9 (0.8) | 4.1 (1.8) | 4.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Score at the End of 5 Minutes of Skin Heating
Description: Verbal pain score measured at one minute intervals during the 5 minute heating of the skin at intervals up to180 minutes after the initiation of the oxytocin infusions, then at 24 hours and 5-7 days after oxytocin infusions. The verbal pain score at the 5 minute measurement is the primary pharmacodynamic outcome for the purpose of modeling the pharmacokinetic-pharmacodynamic relationship. Note that the timing of the primary outcome differs among arms.
  Pain intensity report will be recorded each minute during the heating of the skin to 45 - 47 degrees Celsius . Pain will be determined using a Verbal Pain scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to THE WORST PAIN IMAGINABLE. Heating temperature will be determined according to pain rating during screening visit.
Time Frame: 5-7 days
Population: There was one outlier in the Verbal Pain Score at 20 Minutes group, whose data was not included in the primary analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Verbal Pain Score at 10 Minutes: Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 10, 25, 40, 55, 70, 85, 100, 115, and 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Oxytocin: Intravenous oxytocin
- Verbal Pain Score at 15 Minutes: Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 15, 30, 45, 60, 75, 90, 105, 120, and 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Oxytocin: Intravenous oxytocin
- Verbal Pain Score at 20 Minutes: Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 20, 35, 50, 65, 80, 95, 110, 125, and 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Oxytocin: Intravenous oxytocin
Arm/Group | Verbal Pain Score at 10 Minutes | Verbal Pain Score at 15 Minutes | Verbal Pain Score at 20 Minutes
Number analyzed (Participants) | 8 | 8 | 9
score on a scale
  10 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  10 minutes after starting oxytocin infusion (first arm only) | 3.3 (0.9) |  |
  15 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  15 minutes after starting oxytocin infusion (second arm only) |  | 3.1 (0.9) |
  20 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  20 minutes after starting oxytocin infusion (third arm only) |  |  | 3.4 (1.9)
  25 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  25 minutes after starting oxytocin infusion (first arm only) | 3.1 (1.3) |  |
  30 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  30 minutes after starting oxytocin infusion (second arm only) |  | 3.6 (1.3) |
  35 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  35 minutes after starting oxytocin infusion (third arm only) |  |  | 3.4 (2.2)
  40 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  40 minutes after starting oxytocin infusion (first arm only) | 2.8 (1.0) |  |
  45 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  45 minutes after starting oxytocin infusion (second arm only) |  | 2.4 (1.3) |
  50 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  50 minutes after starting oxytocin infusion (third arm only) |  |  | 3.1 (2.2)
  55 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  55 minutes after starting oxytocin infusion (first arm only) | 3.0 (0.9) |  |
  60 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  60 minutes after starting oxytocin infusion (second arm only) |  | 2.6 (1.0) |
  65 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  65 minutes after starting oxytocin infusion (third arm only) |  |  | 3.2 (2.1)
  70 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  70 minutes after starting oxytocin infusion (first arm only) | 2.3 (1.3) |  |
  75 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  75 minutes after starting oxytocin infusion (second arm only) |  | 2.6 (1.1) |
  80 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  80 minutes after starting oxytocin infusion (third arm only) |  |  | 3.1 (2.2)
  85 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  85 minutes after starting oxytocin infusion (first arm only) | 2.3 (0.9) |  |
  90 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  90 minutes after starting oxytocin infusion (second arm only) |  | 2.1 (0.9) |
  95 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  95 minutes after starting oxytocin infusion (third arm only) |  |  | 3.2 (2.1)
  100 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  100 minutes after starting oxytocin infusion (first arm only) | 2.5 (1.2) |  |
  105 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  105 minutes after starting oxytocin infusion (second arm only) |  | 2.0 (0.8) |
  110 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  110 minutes after starting oxytocin infusion (third arm only) |  |  | 2.9 (2.3)
  115 minutes after starting oxytocin infusion (first arm only): number analyzed (Participants) | 8 | 0 | 0
  115 minutes after starting oxytocin infusion (first arm only) | 2.6 (0.5) |  |
  120 minutes after starting oxytocin infusion (second arm only): number analyzed (Participants) | 0 | 8 | 0
  120 minutes after starting oxytocin infusion (second arm only) |  | 2.1 (1.1) |
  125 minutes after starting oxytocin infusion (third arm only): number analyzed (Participants) | 0 | 0 | 9
  125 minutes after starting oxytocin infusion (third arm only) |  |  | 3.3 (2.5)
  180 minutes after starting oxytocin infusion (all arms) | 2.8 (1.3) | 1.7 (1.7) | 3.5 (2.2)
  24 hours after starting oxytocin infusion (all arms) | 3.0 (1.1) | 2.6 (1.4) | 3.7 (2.0)
  5-7 days after starting oxytocin infusion (all arms) | 3.5 (1.4) | 2.9 (1.1) | 3.7 (1.9)

ADVERSE EVENTS:
Time Frame: 5 to 7 days after oxytocin infusion
Description: On the day of oxytocin infusion, vital signs were recorded at intervals before and up to 180 minutes after beginning the first infusion. Subjects were observed for transient facial flushing and were queried for any adverse events. On visits 24 hr and 5 to 7 days later, subjects were queried regarding any adverse events.
Groups:
- Verbal Pain Score at 10 Minutes: Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 10 minutes after starting the intervention, then every 15 minutes until 115 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Oxytocin: Intravenous oxytocin
- Verbal Pain Score at 15 Minutes: Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 15 minutes after starting the intervention, then every 15 minutes until 120 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Oxytocin: Intravenous oxytocin
- Verbal Pain Score at 20 Minutes: Two 30 minute infusions of oxytocin, 10 IU, will be administered. The second infusion will be given 30 minutes after the completion of the first infusion.
  In this arm the first primary outcome measure (verbal pain report at the end of 5 minutes of skin heating) is obtained at 20 minutes after starting the intervention, then every 15 minutes until 125 minutes and at 180 minutes after starting the intervention. The primary outcome is also measured on separate study visits 24 hours and between 5-7 days after starting the first oxytocin infusion.
  Oxytocin: Intravenous oxytocin
Arm/Group | Verbal Pain Score at 10 Minutes | Verbal Pain Score at 15 Minutes | Verbal Pain Score at 20 Minutes
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 2/8 | 4/8 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verbal Pain Score at 10 Minutes (N=8) | Verbal Pain Score at 15 Minutes (N=8) | Verbal Pain Score at 20 Minutes (N=9)
Flushing (Vascular disorders) | 2 (2) | 4 (4) | 5 (5) — Facial flushing beginning 1 min after starting oxytocin, lasting 1-2 minutes

LIMITATIONS AND CAVEATS:
Analgesic effects from an acute, experimental pain stimulus may not mirror the presence, magnitude and duration of analgesia in clinical settings in the treatment of acute or chronic pain. Additionally, contributions if any, of expectations of efficacy (placebo effect) to pain report were not assessed in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT05929339/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT05929339/ICF_000.pdf